CLINICAL TRIAL: NCT02023606
Title: An Open-Label, Single-Dose, Mass-Balance Study to Assess the Absorption, Metabolism, and Excretion (AME) of [14C] Labeled SPN-810M in Healthy Adult Male Volunteers
Brief Title: Phase I Study to Assess the Absorption, Metabolism, and Excretion of [14C] Labeled SPN-810M
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810P111
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2013-12

CONDITIONS: Impulsive Aggression Comorbid With ADHD
Keywords: Impulsive Aggression; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPN-810M (Experimental): Single dose of 20 mL solution containing 50 mg of SPN-810M and no less than 8.5 MBq (225 µCi) carbon-14 (14C)-SPN-810M, and no more than 11.3 MBq (305 µCi) [14C] SPN-810M.
  Interventions: Drug: SPN-810M

INTERVENTIONS:
Drug: SPN-810M

SUMMARY:
An Open-Label, Single-Dose, Mass-Balance Study to Assess the Absorption, Metabolism, and Excretion of Radio Labeled SPN-810M in Healthy Adult Male Volunteers

ELIGIBILITY:
Key Entry:

1. Healthy males.
2. Aged 30 to 55 years.
3. Considered medically healthy by the Investigator via assessment of physical examination, medical history, clinical laboratory tests, urinalysis, vital signs, and electrocardiogram.
4. Able to voluntarily provide written informed consent to participate in the study.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Urinary and fecal recoveries (mass balance) of total radioactivity. | 10 days post dose.
  C(urine and feces), Ae(urine and feces), CumAe(urine and feces), % Dose(urine and feces), CUM% Dose(urine and feces).

SECONDARY OUTCOMES:
Whole blood and plasma partitioning of total radioactivity. | 10 days post dose.
  To determine whole blood and plasma partitioning of total radioactivity
Pharmacokinetics (PK) of total radioactivity in plasma. | 10 days post dose.
  PK of total radioactivity in plasma (Cmax, Tmax, AUC0-t, AUCinf, Kel, and t1/2).
PK of SPN-810 in plasma. | 10 days post dose.
  PK of SPN-810 in plasma (Cmax, Tmax, AUC0-t, AUCinf, Kel, and t1/2).
PK of the major metabolites of SPN-810 in plasma. | 10 days post dose.
  PK of the major metabolites of SPN-810 in plasma (Cmax, Tmax, AUC0-t, AUCinf, Kel, and t1/2).
Metabolites of SPN-810 in plasma, urine and feces | 10 days post dose.
  To characterize and identify the metabolites of SPN-810 in plasma, urine and feces.
Safety and tolerability of SPN-810. | 10 days post dose.
  To assess the safety and tolerability of SPN-810 by collecting Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Collier, MBChB, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom